CLINICAL TRIAL: NCT00292903
Title: Culturally Relevant Brief Interpersonal Psychotherapy (IPT-B) for Perinatal Depression
Brief Title: Evaluating the Effectiveness of Brief Interpersonal Psychotherapy for Pregnant Women With Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Nancy K. Grote, PhD, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH30915; 5R01MH084897-03 (NIH); DSIR 83-ATSO
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Depression
Keywords: Perinatal Depression; Interpersonal Psychotherapy
MeSH Terms: conditions — Depression | interventions — Therapeutics

ARMS (2):
- A (Experimental)
  Interventions: Behavioral: Brief interpersonal psychotherapy
- B (Active Comparator)
  Interventions: Behavioral: Facilitated referral for treatment as usual

INTERVENTIONS:
Behavioral: Brief interpersonal psychotherapy — IPT-B sessions include evaluation of participants' level of depression, identification of any difficulties or problems that participants may be experiencing, and review of how to manage these problems using skills learned during treatment.
  Arms: A
Behavioral: Facilitated referral for treatment as usual — F-TAU includes providing verbal and written information regarding depressive symptoms and a referral for treatment at a behavioral health clinic.
  Arms: B

SUMMARY:
This study will compare the effectiveness of brief interpersonal psychotherapy versus standard treatment for pregnant women with depression.

DETAILED DESCRIPTION:
Depression is a serious condition affecting millions of people each year. In fact, it is estimated that approximately one in every four women will be treated for a mood disorder, such as depression, at some point in her life. As effective treatment options continue to develop, many women diagnosed with depression are able to resume normal lives and may choose to become pregnant. Also, some women become depressed when pregnant. Interpersonal psychotherapy involves treating psychological difficulties by analyzing problems, talking about possible solutions, and learning more helpful ways of thinking and acting. Brief interpersonal psychotherapy (IPT-B) is a well-tested psychotherapy for depression that has been shortened and modified. The purpose of this study is to evaluate the effectiveness of IPT-B to reduce depressive symptoms in women during pregnancy and to prevent the continuation or recurrence of their depression postpartum.

Participants in this open-label study will be randomly assigned to receive either IPT-B or a facilitated referral for treatment as usual (F-TAU) at an outpatient clinic or community mental health center. Participants assigned to IPT-B will be scheduled to attend eight treatment sessions along with their prenatal clinic visits within a 16-week period. Each treatment session will begin with a brief 1-minute evaluation to assess participants' level of depression and will end with a brief evaluation of the session. Participants will attend follow-up sessions every 2 weeks until 3 months postpartum and then monthly until 6 months postpartum. These sessions will include evaluation of participants' level of depression, identification of any difficulties or problems that participants may be experiencing, and review of how to manage these problems using skills learned during treatment. Participants assigned to receive F-TAU will be provided with verbal and written information regarding their depressive symptoms. They will also receive a referral for treatment at a behavioral health clinic. Participants receiving F-TAU will be assessed via telephone at Weeks 6 and 12. All participants will be assessed via telephone at Months 2 and 6 postpartum to measure their level of depression.

ELIGIBILITY:
Inclusion Criteria:

* Between 8 and 32 weeks of gestation at time of study entry
* A score above 12 on the Edinburgh Postnatal Depression Scale
* Speaks English
* Resides in the Pittsburgh, PA, area
* Access to a household telephone

Exclusion Criteria:

* Currently receiving treatment for depression (i.e., medication or psychotherapy)
* History of a prior manic episode
* Alcohol or drug abuse or dependence within 6 months of study entry
* Psychotic disorder or organic mental disorder
* Suicidal, homicidal, or requires hospitalization
* Severe sexual and/or physical aggression in relationship with partner or husband
* Significant medical illness such as epilepsy, autoimmune disorder, liver dysfunction, or unstable endocrine disease
* Severe cognitive deficits that would prevent treatment with psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2004-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Measured throughout treatment and at Months 2 and 6 postpartum
Treatment attendance | Measured at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K. Grote, PhD, Principal Investigator — University of Pittsburgh, School of Social Work
Locations (1):
- Magee Womens Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Jones KA, Freijah I, Brennan SE, McKenzie JE, Bright TM, Fiolet R, Kamitsis I, Reid C, Davis E, Andrews S, Muzik M, Segal L, Herrman H, Chamberlain C. Interventions from pregnancy to two years after birth for parents experiencing complex post-traumatic stress disorder and/or with childhood experience of maltreatment. Cochrane Database Syst Rev. 2023 May 4;5(5):CD014874. doi: 10.1002/14651858.CD014874.pub2. PMID 37146219